CLINICAL TRIAL: NCT02736890
Title: Subcutaneous Injection of Botulinum Toxin A for At--Level Back Pain in Patients With Spinal Cord Injury
Brief Title: Injecting Botulinum Toxin A Underneath the Skin to Treat Spinal Cord Pain in Patients With Spinal Cord Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding not available to continue
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Thomas N. Bryce, Professor of Rehabilitation Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 14-2212
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Neuropathic Back Pain; Spinal Cord Injury
Keywords: Botulinum Toxin A; Neuropathic pain; Spinal cord injury; Pain management; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia; Agnosia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin A (Active Comparator): Each vial of botulin toxin (100U, BOTOX, Allergan) will be reconstituted with 4ml non-preserved saline solution (0.9%) as recommended by the manufacturer (concentration of 5 units Botulinum Toxin A/0.2ml). Each injection will be 0.2mL (BOTOX, 5 units), administered through a 25 gauge needle. The marked area will have subcutaneous injections, each separated by a radius of 1 cm, from the other injections into the marked area,(maximum of 80 injections, 400 Units).
  Interventions: Drug: Botulinum Toxin A
- Placebo (Placebo Comparator): Placebo consists of 0.9% normal saline. Each injection will be 0.2mL, administered with a 25 gauge needle subcutaneously into the affected area. The marked area will have subcutaneous injections (maximum of 80) each separated from the surrounding ones by a radius of 1 cm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin A — Subjects will receive subcutaneous Botulinum Toxin A injections into the marked painful region. The syringes will be prepared by a third party prior to the injection and the administrator of the procedure will be blinded to syringe content. This physician will be performing the injections under sterile conditions. Local anesthesia, EMLA (lignocaine/prilocaine eutectic mixture) cream, up to 4 grams, will be applied topically for local anesthesia. After 50 minutes, the cream will be cleaned off. Overlying skin will be sterilized with either betadine or alcohol solution.
  Other Names: Botox
  Arms: Botulinum Toxin A
Drug: Placebo — Subjects will receive subcutaneous placebo injections into the marked painful region. The syringes will be prepared by a third party prior to the injection and the administrator of the procedure will be blinded to syringe content. This physician will be performing the injections under sterile conditions. Local anesthesia, EMLA (lignocaine/prilocaine eutectic mixture) cream, up to 4 grams, will be applied topically for local anesthesia. After 50 minutes, the cream will be cleaned off. Overlying skin will be sterilized with either betadine or alcohol solution.
  Arms: Placebo

SUMMARY:
Back pain is a common secondary condition of both acute and chronic spinal cord injury (SCI). Current existing treatment including both pharmacologic and non-pharmacologic are limited by marginal efficacy or intolerable side effects. The purpose of this study is to evaluate the potential of subcutaneous injections of botulinum toxin A to provide pain relief in spinal cord injury patients with back pain near the level of injury in the spine. Botulinum toxin A has been shown in both pre-clinical and clinical studies to help with nerve pain. The researchers propose a double blinded placebo controlled crossover study to study the effects of subcutaneous botulinum injections to at--level SCI back pain in patients with spinal cord injury.

DETAILED DESCRIPTION:
In this study, there will be 2 procedure performed. The first procedure will be named P1 and consists of subcutaneous injection of either placebo or Botulinum Toxin A. The second procedure will be the cross-over procedure named P2. For the cross-over procedure, the subjects who had initially received Botulinum Toxin A will receive placebo and the subjects who had initially received placebo will receive Botulinum Toxin A. This is a Randomized Double-Blinded Placebo Controlled Trial. Recruited subjects will be consented, enrolled and evaluated immediately prior to P1 (or during a visit prior to the visit for P1). After the initial pre-treatment evaluation, subjects will randomly receive either placebo or Botulinum Toxin A subcutaneously (P1). A telephone follow-up (or e-mail follow up) will be performed at 2 weeks and 8 weeks post- P1. An onsite follow up will be performed 4 weeks post P1 and 12 weeks post P1.

Cross-over Study: After the 3rd month on-site evaluation (12 weeks post P1), during the same visit, the subject will proceed to the cross-over study. At this time, the patient will have the option to receive a repeat subcutaneous injection of the cross-over agent. If they desire one, a subcutaneous injection of the cross-over agent will be performed at that same visit. If they wish to defer the repeat injection, they will be contacted and asked every 4 weeks - between 12 weeks and 24 weeks post P1 (no subject will receive P2 after week 24) if they would like to have the subcutaneous injection of the cross-over agent. If they desire one, a repeat injection will be scheduled for the following week.

The rationale for a variable length of time after the initial Botulinum Toxin A/Placebo injection (P1) is to document the variability of individuals' pain response after Botulinum Toxin A. It has been reported in literature, of the subjects that respond to subcutaneous Botulinum Toxin A injections for pain, most will return to their base-line pain score in 12--24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 80 years old
* Diagnosed with traumatic spinal cord injury
* Target pain is considered by the physician as at-level SCI in nature to a high degree of certainty (4 or 5 using a Likert confidence scale ranging from 0-5 where 0 is "purely a guess" and 5 is "absolutely certain")
* Able to give written informed consent
* Target pain that has been continuously present for at least one month
* Target pain is of at least moderate average intensity over the past week, e.g., greater than or equal to 4/10 on a numeric rating scale, the cutoff point for moderate pain in an SCI population.
* Target pain is localized within the dermatome which identifies the NLI or within 3 levels below the NLI
* Subject has been on a stable dose of analgesic mediation (or not on analgesic medication) for at least 3 weeks and is agreeable to remaining on current regimen for the duration of the study (previous prescribed breakthrough analgesics will be allowed)

Exclusion Criteria:

* Pregnancy
* History of intolerance, hypersensitivity or known allergy to botulinum toxin or its preservatives
* History of intolerance, hypersensitivity or known allergy to EMLA cream (lignocaine/prilocaine eutectic mixture) which is used as an analgesic during BoNT injection
* Recent history of administration of botulinum toxin (within previous 6 months)
* Contraindications to botulinum toxin (myasthenia gravis or other disease of the neuromuscular junction)
* Coagulation disorder
* Current infection
* Insufficient command of English to complete self-report instruments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03; Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bryce, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The following will be shared: demographic information, pain response to interventions, adverse events and functional outcomes. The above information will be obtain in the forms of questionnaires and surveys. The data will be available when the study concludes.

REFERENCES:
- [Background] Siddall PJ, McClelland JM, Rutkowski SB, Cousins MJ. A longitudinal study of the prevalence and characteristics of pain in the first 5 years following spinal cord injury. Pain. 2003 Jun;103(3):249-257. doi: 10.1016/S0304-3959(02)00452-9. PMID 12791431
- [Background] Cardenas DD, Bryce TN, Shem K, Richards JS, Elhefni H. Gender and minority differences in the pain experience of people with spinal cord injury. Arch Phys Med Rehabil. 2004 Nov;85(11):1774-81. doi: 10.1016/j.apmr.2004.04.027. PMID 15520972
- [Background] Rintala DH, Loubser PG, Castro J, Hart KA, Fuhrer MJ. Chronic pain in a community-based sample of men with spinal cord injury: prevalence, severity, and relationship with impairment, disability, handicap, and subjective well-being. Arch Phys Med Rehabil. 1998 Jun;79(6):604-14. doi: 10.1016/s0003-9993(98)90032-6. PMID 9630137
- [Background] Jensen MP, Hoffman AJ, Cardenas DD. Chronic pain in individuals with spinal cord injury: a survey and longitudinal study. Spinal Cord. 2005 Dec;43(12):704-12. doi: 10.1038/sj.sc.3101777. PMID 15968299
- [Background] Vogel LC, Krajci KA, Anderson CJ. Adults with pediatric-onset spinal cord injury: part 2: musculoskeletal and neurological complications. J Spinal Cord Med. 2002 Summer;25(2):117-23. doi: 10.1080/10790268.2002.11753611. PMID 12137215
- [Background] McColl MA, Charlifue S, Glass C, Lawson N, Savic G. Aging, gender, and spinal cord injury. Arch Phys Med Rehabil. 2004 Mar;85(3):363-7. doi: 10.1016/j.apmr.2003.06.022. PMID 15031818
- [Background] Knutsdottir S. Spinal cord injuries in Iceland 1973-1989. A follow up study. Paraplegia. 1993 Jan;31(1):68-72. doi: 10.1038/sc.1993.10. PMID 8446450
- [Background] Samuelsson KK. Back pain and spinal Deformity-Common among wheelchair users with spinal cord injuries. Scandinavian journal of occupational therapy. 1996 -01;3(1):28-32.
- [Background] Waisbrod H, Hansen D, Gerbershagen HU. Chronic pain in paraplegics. Neurosurgery. 1984 Dec;15(6):933-4. PMID 6514167
- [Background] Hardcastle P, Bedbrook G, Curtis K. Long-term results of conservative and operative management in complete paraplegics with spinal cord injuries between T10 and L2 with respect to function. Clin Orthop Relat Res. 1987 Nov;(224):88-96. PMID 3665258
- [Background] Walter JS, Sacks J, Othman R, Rankin AZ, Nemchausky B, Chintam R, Wheeler JS. A database of self-reported secondary medical problems among VA spinal cord injury patients: its role in clinical care and management. J Rehabil Res Dev. 2002 Jan-Feb;39(1):53-61. PMID 11926327
- [Background] Rintala DH, Hart KA, Priebe MM. Predicting consistency of pain over a 10-year period in persons with spinal cord injury. J Rehabil Res Dev. 2004 Jan-Feb;41(1):75-88. doi: 10.1682/jrrd.2004.01.0075. PMID 15273900
- [Background] Cardenas DD, Jensen MP. Treatments for chronic pain in persons with spinal cord injury: A survey study. J Spinal Cord Med. 2006;29(2):109-17. doi: 10.1080/10790268.2006.11753864. PMID 16739554
- [Background] Cardenas DD, Warms CA, Turner JA, Marshall H, Brooke MM, Loeser JD. Efficacy of amitriptyline for relief of pain in spinal cord injury: results of a randomized controlled trial. Pain. 2002 Apr;96(3):365-373. doi: 10.1016/S0304-3959(01)00483-3. PMID 11973011
- [Background] Levendoglu F, Ogun CO, Ozerbil O, Ogun TC, Ugurlu H. Gabapentin is a first line drug for the treatment of neuropathic pain in spinal cord injury. Spine (Phila Pa 1976). 2004 Apr 1;29(7):743-51. doi: 10.1097/01.brs.0000112068.16108.3a. PMID 15087796
- [Background] Norrbrink C, Lundeberg T. Tramadol in neuropathic pain after spinal cord injury: a randomized, double-blind, placebo-controlled trial. Clin J Pain. 2009 Mar-Apr;25(3):177-84. doi: 10.1097/AJP.0b013e31818a744d. PMID 19333166
- [Background] Elia AE, Filippini G, Calandrella D, Albanese A. Botulinum neurotoxins for post-stroke spasticity in adults: a systematic review. Mov Disord. 2009 Apr 30;24(6):801-12. doi: 10.1002/mds.22452. PMID 19224614
- [Background] Novak I, Campbell L, Boyce M, Fung VS; Cerebral Palsy Institute. Botulinum toxin assessment, intervention and aftercare for cervical dystonia and other causes of hypertonia of the neck: international consensus statement. Eur J Neurol. 2010 Aug;17 Suppl 2:94-108. doi: 10.1111/j.1468-1331.2010.03130.x. PMID 20633181
- [Background] Sheean G, Lannin NA, Turner-Stokes L, Rawicki B, Snow BJ; Cerebral Palsy Institute. Botulinum toxin assessment, intervention and after-care for upper limb hypertonicity in adults: international consensus statement. Eur J Neurol. 2010 Aug;17 Suppl 2:74-93. doi: 10.1111/j.1468-1331.2010.03129.x. PMID 20633180
- [Background] Olver J, Esquenazi A, Fung VS, Singer BJ, Ward AB; Cerebral Palsy Institute. Botulinum toxin assessment, intervention and aftercare for lower limb disorders of movement and muscle tone in adults: international consensus statement. Eur J Neurol. 2010 Aug;17 Suppl 2:57-73. doi: 10.1111/j.1468-1331.2010.03128.x. PMID 20633179
- [Background] Piovesan EJ, Teive HG, Kowacs PA, Della Coletta MV, Werneck LC, Silberstein SD. An open study of botulinum-A toxin treatment of trigeminal neuralgia. Neurology. 2005 Oct 25;65(8):1306-8. doi: 10.1212/01.wnl.0000180940.98815.74. PMID 16247065
- [Background] Xiao L, Mackey S, Hui H, Xong D, Zhang Q, Zhang D. Subcutaneous injection of botulinum toxin a is beneficial in postherpetic neuralgia. Pain Med. 2010 Dec;11(12):1827-33. doi: 10.1111/j.1526-4637.2010.01003.x. PMID 21134121
- [Background] Wu CJ, Lian YJ, Zheng YK, Zhang HF, Chen Y, Xie NC, Wang LJ. Botulinum toxin type A for the treatment of trigeminal neuralgia: results from a randomized, double-blind, placebo-controlled trial. Cephalalgia. 2012 Apr;32(6):443-50. doi: 10.1177/0333102412441721. Epub 2012 Apr 5. PMID 22492424
- [Background] Yuan RY, Sheu JJ, Yu JM, Chen WT, Tseng IJ, Chang HH, Hu CJ. Botulinum toxin for diabetic neuropathic pain: a randomized double-blind crossover trial. Neurology. 2009 Apr 28;72(17):1473-8. doi: 10.1212/01.wnl.0000345968.05959.cf. Epub 2009 Feb 25. PMID 19246421
- [Background] Jabbari B, Maher N, Difazio MP. Botulinum toxin a improved burning pain and allodynia in two patients with spinal cord pathology. Pain Med. 2003 Jun;4(2):206-10. doi: 10.1046/j.1526-4637.2003.03013.x. PMID 12873271
- [Background] Bryce TN, Budh CN, Cardenas DD, Dijkers M, Felix ER, Finnerup NB, Kennedy P, Lundeberg T, Richards JS, Rintala DH, Siddall P, Widerstrom-Noga E. Pain after spinal cord injury: an evidence-based review for clinical practice and research. Report of the National Institute on Disability and Rehabilitation Research Spinal Cord Injury Measures meeting. J Spinal Cord Med. 2007;30(5):421-40. doi: 10.1080/10790268.2007.11753405. PMID 18092558
- [Background] Bryce TN, Biering-Sorensen F, Finnerup NB, Cardenas DD, Defrin R, Ivan E, Lundeberg T, Norrbrink C, Richards JS, Siddall P, Stripling T, Treede RD, Waxman SG, Widerstrom-Noga E, Yezierski RP, Dijkers M. International Spinal Cord Injury Pain (ISCIP) Classification: Part 2. Initial validation using vignettes. Spinal Cord. 2012 Jun;50(6):404-12. doi: 10.1038/sc.2012.2. Epub 2012 Feb 7. PMID 22310319
- [Background] Bryce TN, Ragnarsson KT. Pain after spinal cord injury. Phys Med Rehabil Clin N Am. 2000 Feb;11(1):157-68. PMID 10680163
- [Background] Vranken JH, Hollmann MW, van der Vegt MH, Kruis MR, Heesen M, Vos K, Pijl AJ, Dijkgraaf MGW. Duloxetine in patients with central neuropathic pain caused by spinal cord injury or stroke: a randomized, double-blind, placebo-controlled trial. Pain. 2011 Feb;152(2):267-273. doi: 10.1016/j.pain.2010.09.005. PMID 21078545
- [Background] Lis AM, Black KM, Korn H, Nordin M. Association between sitting and occupational LBP. Eur Spine J. 2007 Feb;16(2):283-98. doi: 10.1007/s00586-006-0143-7. Epub 2006 May 31. PMID 16736200
- [Background] Van Nieuwenhuyse A, Fatkhutdinova L, Verbeke G, Pirenne D, Johannik K, Somville PR, Mairiaux P, Moens GF, Masschelein R. Risk factors for first-ever low back pain among workers in their first employment. Occup Med (Lond). 2004 Dec;54(8):513-9. doi: 10.1093/occmed/kqh091. Epub 2004 Sep 22. PMID 15385649
- [Background] Adams MA, McNally DS, Chinn H, Dolan P. The clinical biomechanics award paper 1993 Posture and the compressive strength of the lumbar spine. Clin Biomech (Bristol). 1994 Jan;9(1):5-14. doi: 10.1016/0268-0033(94)90052-3. PMID 23916072
- [Background] Panjabi MM, Andersson GB, Jorneus L, Hult E, Mattsson L. In vivo measurements of spinal column vibrations. J Bone Joint Surg Am. 1986 Jun;68(5):695-702. PMID 3722226
- [Background] Scannell JP, McGill SM. Lumbar posture--should it, and can it, be modified? A study of passive tissue stiffness and lumbar position during activities of daily living. Phys Ther. 2003 Oct;83(10):907-17. PMID 14519062
- [Background] Claus AP, Hides JA, Moseley GL, Hodges PW. Is 'ideal' sitting posture real? Measurement of spinal curves in four sitting postures. Man Ther. 2009 Aug;14(4):404-8. doi: 10.1016/j.math.2008.06.001. Epub 2008 Sep 14. PMID 18793867
- [Background] Dunk NM, Kedgley AE, Jenkyn TR, Callaghan JP. Evidence of a pelvis-driven flexion pattern: are the joints of the lower lumbar spine fully flexed in seated postures? Clin Biomech (Bristol). 2009 Feb;24(2):164-8. doi: 10.1016/j.clinbiomech.2008.12.003. Epub 2009 Jan 12. PMID 19138810
- [Background] De Carvalho DE, Soave D, Ross K, Callaghan JP. Lumbar spine and pelvic posture between standing and sitting: a radiologic investigation including reliability and repeatability of the lumbar lordosis measure. J Manipulative Physiol Ther. 2010 Jan;33(1):48-55. doi: 10.1016/j.jmpt.2009.11.008. PMID 20114100
- [Background] Dolan P, Adams MA, Hutton WC. Commonly adopted postures and their effect on the lumbar spine. Spine (Phila Pa 1976). 1988 Feb;13(2):197-201. doi: 10.1097/00007632-198802000-00012. PMID 3406840
- [Background] Lord MJ, Small JM, Dinsay JM, Watkins RG. Lumbar lordosis. Effects of sitting and standing. Spine (Phila Pa 1976). 1997 Nov 1;22(21):2571-4. doi: 10.1097/00007632-199711010-00020. PMID 9383867
- [Background] Callaghan JP, McGill SM. Low back joint loading and kinematics during standing and unsupported sitting. Ergonomics. 2001 Feb 20;44(3):280-94. doi: 10.1080/00140130118276. PMID 11219760
- [Background] Harrison DD, Harrison SO, Croft AC, Harrison DE, Troyanovich SJ. Sitting biomechanics part I: review of the literature. J Manipulative Physiol Ther. 1999 Nov-Dec;22(9):594-609. doi: 10.1016/s0161-4754(99)70020-5. PMID 10626703
- [Background] Hedman TP, Fernie GR. Mechanical response of the lumbar spine to seated postural loads. Spine (Phila Pa 1976). 1997 Apr 1;22(7):734-43. doi: 10.1097/00007632-199704010-00004. PMID 9106313
- [Background] Reeve A, Dilley A. Effects of posture on the thickness of transversus abdominis in pain-free subjects. Man Ther. 2009 Dec;14(6):679-84. doi: 10.1016/j.math.2009.02.008. Epub 2009 May 14. PMID 19443261
- [Background] Claus AP, Hides JA, Moseley GL, Hodges PW. Different ways to balance the spine: subtle changes in sagittal spinal curves affect regional muscle activity. Spine (Phila Pa 1976). 2009 Mar 15;34(6):E208-14. doi: 10.1097/BRS.0b013e3181908ead. PMID 19282726
- [Background] O'Sullivan PB, Dankaerts W, Burnett AF, Farrell GT, Jefford E, Naylor CS, O'Sullivan KJ. Effect of different upright sitting postures on spinal-pelvic curvature and trunk muscle activation in a pain-free population. Spine (Phila Pa 1976). 2006 Sep 1;31(19):E707-12. doi: 10.1097/01.brs.0000234735.98075.50. PMID 16946644
- [Background] Francisco GE, Tan H, Green M. Do botulinum toxins have a role in the management of neuropathic pain?: a focused review. Am J Phys Med Rehabil. 2012 Oct;91(10):899-909. doi: 10.1097/PHM.0b013e31825a134b. PMID 22660369
- [Background] Lu DW, Lippitz J. Complications of botulinum neurotoxin. Dis Mon. 2009 Apr;55(4):198-211. doi: 10.1016/j.disamonth.2009.01.001. No abstract available. PMID 19286054
- [Background] Argoff CE. A focused review on the use of botulinum toxins for neuropathic pain. Clin J Pain. 2002 Nov-Dec;18(6 Suppl):S177-81. doi: 10.1097/00002508-200211001-00010. PMID 12569966
- [Background] Matak I, Bach-Rojecky L, Filipovic B, Lackovic Z. Behavioral and immunohistochemical evidence for central antinociceptive activity of botulinum toxin A. Neuroscience. 2011 Jul 14;186:201-7. doi: 10.1016/j.neuroscience.2011.04.026. Epub 2011 Apr 20. PMID 21539899
- [Background] Foster L, Clapp L, Erickson M, Jabbari B. Botulinum toxin A and chronic low back pain: a randomized, double-blind study. Neurology. 2001 May 22;56(10):1290-3. doi: 10.1212/wnl.56.10.1290. PMID 11376175
- [Background] Apalla Z, Sotiriou E, Lallas A, Lazaridou E, Ioannides D. Botulinum toxin A in postherpetic neuralgia: a parallel, randomized, double-blind, single-dose, placebo-controlled trial. Clin J Pain. 2013 Oct;29(10):857-64. doi: 10.1097/AJP.0b013e31827a72d2. PMID 23370074
- [Background] Ranoux D, Attal N, Morain F, Bouhassira D. Botulinum toxin type A induces direct analgesic effects in chronic neuropathic pain. Ann Neurol. 2008 Sep;64(3):274-83. doi: 10.1002/ana.21427. PMID 18546285
- [Background] Bach-Rojecky L, Salkovic-Petrisic M, Lackovic Z. Botulinum toxin type A reduces pain supersensitivity in experimental diabetic neuropathy: bilateral effect after unilateral injection. Eur J Pharmacol. 2010 May 10;633(1-3):10-4. doi: 10.1016/j.ejphar.2010.01.020. Epub 2010 Feb 1. PMID 20123097
- [Background] Bach-Rojecky L, Lackovic Z. Central origin of the antinociceptive action of botulinum toxin type A. Pharmacol Biochem Behav. 2009 Dec;94(2):234-8. doi: 10.1016/j.pbb.2009.08.012. Epub 2009 Sep 2. PMID 19732788
- [Background] Kharkar S, Ambady P, Venkatesh Y, Schwartzman RJ. Intramuscular botulinum toxin in complex regional pain syndrome: case series and literature review. Pain Physician. 2011 Sep-Oct;14(5):419-24. PMID 21927045
- [Background] Birthi P, Sloan P, Salles S. Subcutaneous botulinum toxin A for the treatment of refractory complex regional pain syndrome. PM R. 2012 Jun;4(6):446-9. doi: 10.1016/j.pmrj.2011.12.010. No abstract available. PMID 22732156
- [Background] Fabregat G, Asensio-Samper JM, Palmisani S, Villanueva-Perez VL, De Andres J. Subcutaneous botulinum toxin for chronic post-thoracotomy pain. Pain Pract. 2013 Mar;13(3):231-4. doi: 10.1111/j.1533-2500.2012.00569.x. Epub 2012 Jun 21. PMID 22716282
- [Background] Zhang T, Adatia A, Zarin W, Moitri M, Vijenthira A, Chu R, Thabane L, Kean W. The efficacy of botulinum toxin type A in managing chronic musculoskeletal pain: a systematic review and meta analysis. Inflammopharmacology. 2011 Feb;19(1):21-34. doi: 10.1007/s10787-010-0069-x. Epub 2010 Nov 13. PMID 21076878
- [Background] Argoff C. The emerging use of botulinum toxins for the treatment of neuropathic pain. Pain Med. 2010 Dec;11(12):1750-2. doi: 10.1111/j.1526-4637.2010.00997.x. No abstract available. PMID 21134116
- [Background] Lew HL, Lee EH, Castaneda A, Klima R, Date E. Therapeutic use of botulinum toxin type A in treating neck and upper-back pain of myofascial origin: a pilot study. Arch Phys Med Rehabil. 2008 Jan;89(1):75-80. doi: 10.1016/j.apmr.2007.08.133. PMID 18164334
- [Background] Jabbari B, Machado D. Treatment of refractory pain with botulinum toxins--an evidence-based review. Pain Med. 2011 Nov;12(11):1594-606. doi: 10.1111/j.1526-4637.2011.01245.x. Epub 2011 Sep 29. PMID 21958302
- [Background] Jabbari B, Ney J, Sichani A, Monacci W, Foster L, Difazio M. Treatment of refractory, chronic low back pain with botulinum neurotoxin A: an open-label, pilot study. Pain Med. 2006 May-Jun;7(3):260-4. doi: 10.1111/j.1526-4637.2006.00147.x. PMID 16712627
- [Background] McMahon HT, Foran P, Dolly JO, Verhage M, Wiegant VM, Nicholls DG. Tetanus toxin and botulinum toxins type A and B inhibit glutamate, gamma-aminobutyric acid, aspartate, and met-enkephalin release from synaptosomes. Clues to the locus of action. J Biol Chem. 1992 Oct 25;267(30):21338-43. PMID 1356988
- [Background] Welch MJ, Purkiss JR, Foster KA. Sensitivity of embryonic rat dorsal root ganglia neurons to Clostridium botulinum neurotoxins. Toxicon. 2000 Feb;38(2):245-58. doi: 10.1016/s0041-0101(99)00153-1. PMID 10665805
- [Background] Durham PL, Cady R, Cady R. Regulation of calcitonin gene-related peptide secretion from trigeminal nerve cells by botulinum toxin type A: implications for migraine therapy. Headache. 2004 Jan;44(1):35-42; discussion 42-3. doi: 10.1111/j.1526-4610.2004.04007.x. PMID 14979881
- [Background] Meng J, Wang J, Lawrence G, Dolly JO. Synaptobrevin I mediates exocytosis of CGRP from sensory neurons and inhibition by botulinum toxins reflects their anti-nociceptive potential. J Cell Sci. 2007 Aug 15;120(Pt 16):2864-74. doi: 10.1242/jcs.012211. Epub 2007 Jul 31. PMID 17666428
- [Background] Planells-Cases R, Garcia-Sanz N, Morenilla-Palao C, Ferrer-Montiel A. Functional aspects and mechanisms of TRPV1 involvement in neurogenic inflammation that leads to thermal hyperalgesia. Pflugers Arch. 2005 Oct;451(1):151-9. doi: 10.1007/s00424-005-1423-5. Epub 2005 May 21. PMID 15909179
- [Background] Morenilla-Palao C, Planells-Cases R, Garcia-Sanz N, Ferrer-Montiel A. Regulated exocytosis contributes to protein kinase C potentiation of vanilloid receptor activity. J Biol Chem. 2004 Jun 11;279(24):25665-72. doi: 10.1074/jbc.M311515200. Epub 2004 Apr 5. PMID 15066994
- [Background] Antonucci F, Rossi C, Gianfranceschi L, Rossetto O, Caleo M. Long-distance retrograde effects of botulinum neurotoxin A. J Neurosci. 2008 Apr 2;28(14):3689-96. doi: 10.1523/JNEUROSCI.0375-08.2008. PMID 18385327
- [Background] Restani L, Antonucci F, Gianfranceschi L, Rossi C, Rossetto O, Caleo M. Evidence for anterograde transport and transcytosis of botulinum neurotoxin A (BoNT/A). J Neurosci. 2011 Nov 2;31(44):15650-9. doi: 10.1523/JNEUROSCI.2618-11.2011. PMID 22049408
- [Background] Naumann M, Jankovic J. Safety of botulinum toxin type A: a systematic review and meta-analysis. Curr Med Res Opin. 2004 Jul;20(7):981-90. doi: 10.1185/030079904125003962. PMID 15265242
- [Background] Naumann M, Albanese A, Heinen F, Molenaers G, Relja M. Safety and efficacy of botulinum toxin type A following long-term use. Eur J Neurol. 2006 Dec;13 Suppl 4:35-40. doi: 10.1111/j.1468-1331.2006.01652.x. PMID 17112348
- [Background] Li M, Goldberger BA, Hopkins C. Fatal case of BOTOX-related anaphylaxis? J Forensic Sci. 2005 Jan;50(1):169-72. PMID 15831014
- [Background] Forchheimer MB, Richards JS, Chiodo AE, Bryce TN, Dyson-Hudson TA. Cut point determination in the measurement of pain and its relationship to psychosocial and functional measures after traumatic spinal cord injury: a retrospective model spinal cord injury system analysis. Arch Phys Med Rehabil. 2011 Mar;92(3):419-24. doi: 10.1016/j.apmr.2010.08.029. PMID 21353824
- [Background] Hanley MA, Jensen MP, Ehde DM, Robinson LR, Cardenas DD, Turner JA, Smith DG. Clinically significant change in pain intensity ratings in persons with spinal cord injury or amputation. Clin J Pain. 2006 Jan;22(1):25-31. doi: 10.1097/01.ajp.0000148628.69627.82. PMID 16340590
- [Background] BEECHER HK. The powerful placebo. J Am Med Assoc. 1955 Dec 24;159(17):1602-6. doi: 10.1001/jama.1955.02960340022006. No abstract available. PMID 13271123
- [Background] Widerstrom-Noga E, Biering-Sorensen F, Bryce T, Cardenas DD, Finnerup NB, Jensen MP, Richards JS, Siddall PJ. The international spinal cord injury pain basic data set. Spinal Cord. 2008 Dec;46(12):818-23. doi: 10.1038/sc.2008.64. Epub 2008 Jun 3. PMID 18521092
- [Background] Jensen MP, Widerstrom-Noga E, Richards JS, Finnerup NB, Biering-Sorensen F, Cardenas DD. Reliability and validity of the International Spinal Cord Injury Basic Pain Data Set items as self-report measures. Spinal Cord. 2010 Mar;48(3):230-8. doi: 10.1038/sc.2009.112. Epub 2009 Sep 29. PMID 19786975
- [Background] Ruta DA, Garratt AM, Leng M, Russell IT, MacDonald LM. A new approach to the measurement of quality of life. The Patient-Generated Index. Med Care. 1994 Nov;32(11):1109-26. doi: 10.1097/00005650-199411000-00004. PMID 7967852
- [Background] Ruta DA, Garratt AM, Russell IT. Patient centred assessment of quality of life for patients with four common conditions. Qual Health Care. 1999 Mar;8(1):22-9. doi: 10.1136/qshc.8.1.22. PMID 10557665
- [Background] Tugwell P, Bombardier C, Buchanan WW, Goldsmith CH, Grace E, Hanna B. The MACTAR Patient Preference Disability Questionnaire--an individualized functional priority approach for assessing improvement in physical disability in clinical trials in rheumatoid arthritis. J Rheumatol. 1987 Jun;14(3):446-51. PMID 3305931
- [Background] Wright JG, Young NL. The patient-specific index: asking patients what they want. J Bone Joint Surg Am. 1997 Jul;79(7):974-83. doi: 10.2106/00004623-199707000-00003. PMID 9234873

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin A Then Placebo: Injection 0.2mL (BOTOX, 5 units), with maximum of 80 injections, 400 Units for 12 weeks, then Placebo 0.2mL of 0.9% normal saline for 12 weeks.
- Placebo Then Botulinum Toxin A: Placebo 0.2mL of 0.9% normal saline for 12 weeks, then Injection 0.2mL (BOTOX, 5 units), with maximum of 80 injections, 400 Units for 12 weeks.
Period: First 12 Weeks
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0
Period: Crossover Next 12 Weeks
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Started | 5 | 3
Completed | 3 | 1
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (7.02) | 36.7 (4.04) | 45.4 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 2 | 1 | 3
  Black or African American | 2 | 0 | 2
  White | 1 | 1 | 2
  Unknown/Not reported | 0 | 1 | 1
DN4 screen (neuropathic >4) [Count of Participants; unit: Participants] — Number of participants scoring >4 on each question on the DN4. Douleur Neuropathique en 4 Questions (DN4) is a screening tool for neuropathic pain consisting of interview questions (DN4-interview) and physical tests. DN4 consists of 7 items related to symptoms and 3 related to clinical examination, total score from 0-10, with higher score indicating more symptom.
  Participants
    Burning | 4 | 2 | 6
    Painful cold | 1 | 2 | 3
    Electric shock | 3 | 2 | 5
    Tingling | 4 | 3 | 7
    Pins and needles | 5 | 3 | 8
    Numbness | 4 | 1 | 5
    Itching | 1 | 2 | 3
    Hypoesthesia to touch | 2 | 1 | 3
    Hypoesthesia to prick | 1 | 1 | 2
    Brushing | 2 | 1 | 3
SCIPI screen (neuropathic >=3) [Count of Participants; unit: Participants] — Number of participants scoring >=3 on each item on the SCIPI. Spinal Cord Injury Pain Instrument is a 7 item instrument, total score from 0-7 with higher score indicating more pain.
  Participants
    Electric shock | 3 | 2 | 5
    Pins and needles | 5 | 3 | 8
    Burning or freezing | 2 | 2 | 4
    Sensitive | 1 | 3 | 4
    Unchanged with movement | 5 | 3 | 8
    All the time when awake | 5 | 3 | 8
    No feeling in area | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: Participant rated pain intensity from 0-10, with higher score indicating more pain
Time Frame: up to 12 weeks post-injection, for a total of 24 weeks from baseline
Population: only those who completed crossover were included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Number analyzed (Participants) | 5 | 3
score on a scale
  baseline | 7.6 (1.5) | 8 (0)
  2 week post injection | 6.4 (0.9) | 8 (0)
  4 week post injection | 5.6 (1.7) | 8 (0)
  8 week post injection | 5.6 (2.6) | 8 (0)
  12 week post injection | 5.6 (3.3) | 8 (0)
  crossover 2 week follow up: number analyzed (Participants) | 3 | 1
  crossover 2 week follow up | 8 (0) | 5 (0)
  crossover 4 week follow up: number analyzed (Participants) | 3 | 1
  crossover 4 week follow up | 8 (0) | 5 (0)
  crossover 8 week follow up: number analyzed (Participants) | 3 | 1
  crossover 8 week follow up | 6.7 (1.5) | 6 (0)
  crossover 12 week follow up: number analyzed (Participants) | 3 | 1
  crossover 12 week follow up | 8 (1) | 7 (0)

2. Secondary Outcome: 7-Point Guy/Farrar Patient Global Impression of Change (PGIC)
Description: Mean change from baseline. Participants are asked "Taking into account your pain level and how it affects your life, are you feeling better, the same or worse than when you started treatment?" and then to quantify the magnitude of the change. with the 7-Point guy Farrar which measures the global treatment effect from with scale from 0 to 6, higher score indicates worse outcomes.
Time Frame: up to 12 weeks post-injection, for a total of 24 weeks from baseline
Population: only those who completed crossover were included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Number analyzed (Participants) | 5 | 3
score on a scale
  2 week post injection | 2.2 (2.2) | 0.3 (0.6)
  4 week post injection | 2.4 (1.5) | 0.3 (0.6)
  8 week post injection | 2 (1.6) | 0 (0)
  12 week post injection | 2 (1.9) | 0 (0)
  crossover 2 week follow up: number analyzed (Participants) | 3 | 1
  crossover 2 week follow up | 0 (0) | 5 (0)
  crossover 4 week follow up: number analyzed (Participants) | 3 | 1
  crossover 4 week follow up | 0 (0) | 5 (0)
  crossover 8 week follow up: number analyzed (Participants) | 3 | 1
  crossover 8 week follow up | 0 (0) | 3 (0)
  crossover 12 week follow up: number analyzed (Participants) | 3 | 1
  crossover 12 week follow up | 0 (0) | 1 (0)

3. Secondary Outcome: International Basic Pain Dataset - Pain Affecting Day-to-day Activities
Description: The International Basic Pain Dataset is an assessment tool which includes several components including: location of pain, temporal qualities of the pain, type of pain, pain interference measures of activity, sleep, and mood. It has been shown to be valid in an interview/self -report format. The pain affecting day-to-day activities subset of the dataset is scored is from 0 to 10, with higher score indicating less favorable outcomes.
Time Frame: up to 12 weeks post-injection, for a total of 24 weeks from baseline
Population: only those who completed crossover were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Number analyzed (Participants) | 5 | 3
units on a scale
  Baseline | 4.2 (4.1) | 5.3 (4.6)
  2 week post injection | 5.4 (1.5) | 2.7 (4.6)
  4 week post injection | 5 (1.2) | 2.7 (4.6)
  8 week post injection | 5 (1.6) | 2.7 (4.6)
  12 week post injection | 4.8 (2.0) | 2.7 (4.6)
  crossover 2 week follow up: number analyzed (Participants) | 3 | 1
  crossover 2 week follow up | 7 (1.7) | 2 (0)
  crossover 4 week follow up: number analyzed (Participants) | 3 | 1
  crossover 4 week follow up | 6.7 (2.3) | 3 (0)
  crossover 8 week follow up: number analyzed (Participants) | 3 | 1
  crossover 8 week follow up | 7 (2.6) | 4 (0)
  crossover 12 week follow up: number analyzed (Participants) | 3 | 1
  crossover 12 week follow up | 6.7 (3.2) | 5 (0)

4. Secondary Outcome: International Basic Pain Dataset - Pain Affecting Mood
Description: The International Basic Pain Dataset is an assessment tool which includes several components including: location of pain, temporal qualities of the pain, type of pain, pain interference measures of activity, sleep, and mood. It has been shown to be valid in an interview/self -report format. The pain affecting mood subset of the dataset is scored is from 0 to 10, with higher score indicating less favorable outcomes.
Time Frame: up to 12 weeks post-injection, for a total of 24 weeks from baseline
Population: only those who completed crossover were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Number analyzed (Participants) | 5 | 3
units on a scale
  Baseline | 5.6 (3.5) | 5.7 (4.9)
  2 week post injection | 6.6 (2.3) | 2.7 (4.6)
  4 week post injection | 5.8 (1.5) | 2.7 (4.6)
  8 week post injection | 5.2 (0.8) | 4.3 (4.5)
  12 week post injection | 5.6 (1.8) | 5.7 (4.9)
  crossover 2 week follow up: number analyzed (Participants) | 3 | 1
  crossover 2 week follow up | 7 (1.7) | 2 (0)
  crossover 4 week follow up: number analyzed (Participants) | 3 | 1
  crossover 4 week follow up | 7 (1.7) | 3 (0)
  crossover 8 week follow up: number analyzed (Participants) | 3 | 1
  crossover 8 week follow up | 7.3 (2.1) | 4 (0)
  crossover 12 week follow up: number analyzed (Participants) | 3 | 1
  crossover 12 week follow up | 6.7 (3.2) | 7 (0)

5. Secondary Outcome: International Basic Pain Dataset - Pain Affecting Sleep
Description: The International Basic Pain Dataset is an assessment tool which includes several components including: location of pain, temporal qualities of the pain, type of pain, pain interference measures of activity, sleep, and mood. It has been shown to be valid in an interview/self -report format. The pain affecting sleep subset of the dataset is scored is from 0 to 10, with higher score indicating less favorable outcomes.
Time Frame: up to 12 weeks post-injection, for a total of 24 weeks from baseline
Population: only those who completed crossover were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Number analyzed (Participants) | 5 | 3
units on a scale
  Baseline | 5.8 (3.8) | 6.7 (2.3)
  2 week post injection | 4.6 (3.6) | 4.7 (3.1)
  4 week post injection | 5 (2.3) | 3.3 (4.2)
  8 week post injection | 6 (1.6) | 6 (2.0)
  12 week post injection | 6.2 (2.2) | 6.7 (2.3)
  crossover 2 week follow up: number analyzed (Participants) | 3 | 1
  crossover 2 week follow up | 8 (0) | 1 (0)
  crossover 4 week follow up: number analyzed (Participants) | 3 | 1
  crossover 4 week follow up | 8 (0) | 3 (0)
  crossover 8 week follow up: number analyzed (Participants) | 3 | 1
  crossover 8 week follow up | 8 (0) | 4 (0)
  crossover 12 week follow up: number analyzed (Participants) | 3 | 1
  crossover 12 week follow up | 7.3 (2.1) | 5 (0)

6. Secondary Outcome: Static Mechanical Allodynia Testing
Description: Mechanical allodynia is a characteristic of evoked pain in subjects with neuropathic pain. Static allodynia to mechanical stimuli will be defined as a sensation of pain evoked by the pressure of the end of a wooden stick. The end of a wooden stick will touch the affected region with enough pressure to indent the skin, for 10 seconds. Afterwards, the subject will be asked to rate the perceived pain on an 11-point NRS.
Time Frame: up to 12 weeks post-injection, for a total of 24 weeks from baseline
Population: Data initially collected incorrectly, then data not collected.
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Dynamic Mechanical Allodynia Testing
Description: Dynamic allodynia will be tested by stroking the affected region gently with a cotton swab, 4 times at a rate of 3-5cm per second over an area of 5cm. If there is an evoked clear sensation of pain, the subject is asked to rate the intensity of dynamic allodynia using the 11-point NRS. The region of static and dynamic allodynia, if present, will be marked and recorded
Time Frame: up to 12 weeks post-injection, for a total of 24 weeks from baseline
Population: Data initially collected incorrectly, then data not collected.
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patient-generated Index (PGI)
Description: PGI measures activity affected by pain. Full score is 0 to 10000, with higher score indicating better function
Time Frame: up to 12 weeks post-injection, for a total of 24 weeks from baseline
Population: only those who completed crossover were included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin A Then Placebo | Placebo Then Botulinum Toxin A
Number analyzed (Participants) | 5 | 3
score on a scale
  Baseline | 4250 (1885.5) | 1500 (1802.8)
  2 week post injection | 5240 (1892.9) | 1550 (1789.6)
  4 week post injection | 5219 (2130.8) | 1825 (2439.5)
  8 week post injection | 3725 (1492.5) | 2800 (2498.0)
  12 week post injection | 4330 (2038.9) | 1800 (2545.6)
  crossover 2 week follow up: number analyzed (Participants) | 3 | 1
  crossover 2 week follow up | 3333.3 (763.8) | 3500 (0)
  crossover 4 week follow up: number analyzed (Participants) | 3 | 1
  crossover 4 week follow up | 3333.3 (763.8) | 3750 (0)
  crossover 8 week follow up: number analyzed (Participants) | 3 | 1
  crossover 8 week follow up | 3333.3 (763.8) | 3000 (0)
  crossover 12 week follow up: number analyzed (Participants) | 3 | 1
  crossover 12 week follow up | 3333.3 (763.8) | 1500 (0)

ADVERSE EVENTS:
Time Frame: 24 weeks post injection
Groups:
- Botulinum Toxin A: Injection 0.2mL (BOTOX, 5 units), with maximum of 80 injections, 400 Units for 12 weeks
- Placebo: Placebo 0.2mL of 0.9% normal saline for 12 weeks
Arm/Group | Botulinum Toxin A | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin A (N=8) | Placebo (N=8)
thrombosed IVCF (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin A (N=8) | Placebo (N=8)
fever (Infections and infestations) | 1 | 0 — Not close to time of injection

LIMITATIONS AND CAVEATS:
Target number of participants needed to achieve target power and statistically reliable results not reached. Unsuccessful questionnaires post injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Recipient will have all rights to data resulting from the Study; provided, however, at least 30 calendar days prior to any submission...Recipient shall provide Allergan a copy of the proposed publication for review. Recipient agrees to delay submission for an additional 30 calendar days to allow Allergan the right to a) address any factual inaccuracies with the publisher as it relates to any Allergan materials or b) request redaction of information that Allergan deems confidential or proprietary

DOCUMENTS (2):
  • Study Protocol (2015-12-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT02736890/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT02736890/SAP_001.pdf